CLINICAL TRIAL: NCT02817139
Title: Transcranial Direct Current Simulation Over Primary Motor vs Prefrontal Cortex in Chronic Migraine: a Pilot Randomized Controlled Trial
Brief Title: Transcranial Direct Current Simulation in Chronic Migraine
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Suellen Marinho Andrade, Professor, Federal University of Paraíba
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: migraine
Record Dates: First submitted 2016-06-22; First posted 2016-06-29 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- active tDCS over primary motor cortex (Active Comparator): Duration: 20 minutes; Intensity: 2 mA; Placement: left primary motor cortex.
  Interventions: Device: TDCS
- active tDCS over prefrontal cortex (Experimental): Duration: 20 minutes; Intensity: 2 mA; Placement: left prefrontal cortex.
  Interventions: Device: TDCS
- sham tDCS over primary motor cortex (Placebo Comparator): Duration: 20 minutes; The procedure is the same as for active tDCS, but the in the placebo tDCS the stimulation is non-active / sham; Placement: left primary motor cortex.
  Interventions: Device: TDCS

INTERVENTIONS:
Device: TDCS
  Other Names: Transcranial Direct Current Stimulation

SUMMARY:
This study is a pilot, double-blind, placebo-controlled, randomized trial aiming to compare the effects of transcranial direct current stimulation in Chronic Migraine.

DETAILED DESCRIPTION:
The patients will be randomized into 1 of 3 groups: active tDCS over primary motor cortex, active tDCS over prefrontal cortex, sham tDCS. Each group will receive treatment for 20 minutes a day, 3 days a week for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* patients with a clinical diagnosis of chronic migraine according to the International Classification of Headaches Disorders (ICHD-3 beta) of the International Headache Society, with an established headache history occurring on 15 or more days per month-however, for at least 1 year, instead of only 3 months, as defined in the International Headache Society (IHS) guidelines.

Exclusion Criteria:

* headache attributable to some pathological condition, associated neurologic or neuropsychiatric disease, use of central nervous system modulating drugs, pregnancy, metallic head implants, and use of a cardiac pacemaker.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life associate to migraine assessed on the Headache Impact Test-6 (HIT-6) | Baseline (week 1) and Endpoint (week 4)

SECONDARY OUTCOMES:
Change in pain assessed on the Visual Analogue Scale (VAS) | Baseline (week 1) and Endpoint (week 4)
Change in quality of life assessed on the Medical Outcomes Study 36 - Item Short - Form Health Survey(SF-36) | Baseline (week 1) and and Endpoint (week 4)
Side Effects Questionnaire | From date of first neurostimulation until the date of last neurostimulation, , assessed up to 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Suellen Andrade, João Pessoa, Paraíba, Brazil